CLINICAL TRIAL: NCT02800746
Title: Preoperative Intravenous Iron Supplementation on Postoperative Hematocrit and Intraoperative Transfusion Amount in Prognathic Surgery
Brief Title: Intravenous Iron Pre-treatment in Prognathic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Tae-Yop Kim, MD PhD, Professor, Konkuk University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KUH1160000
Record Dates: First submitted 2016-06-11; First posted 2016-06-15 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Prognathic Surgery
Keywords: Prognathic surgery; intravenous iron
MeSH Terms: interventions — ferric carboxymaltose; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Ferric carboxymaltose
  Interventions: Drug: Ferric carboxymaltose
- Control Group (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ferric carboxymaltose — Ferric carboxymaltose 15 mg/kg mg is intravenously administered on 7-10 day before surgery.
  Arms: Experimental group
Drug: Placebo — normal saline 100 ml is intravenously administered on 7-10 day before surgery
  Other Names: normal saline
  Arms: Control Group

SUMMARY:
The objective of the present study is to determine the impact of preoperative IV-iron (ferric carboxy maltose) supplementation on postoperative hematocrit values and allogenic blood transfusion amount in patients undergoing elective prognathic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with prognathism in undergoing elective prognathic surgery
* Patients provided a written informed consent.
* Patients with s-ferritin < 300 mg/dl (male) or 200 mg/dl (female)
* Patients with preoperative Hematocrit > 39% (male) and > 36% 9female)serum hemoglobin >13 g/dL (male) and >12 g/dL (female)

Exclusion Criteria:

* Patients with history of anaphylaxis, iron overload, active infection.
* Patients with endocrine disease
* Patients received or receiving intraoperative and preoperative blood salvaged, allogenic blood transfusion, anti-fibrinolytic agents or recombinant human erythropoietin, or undergoing acute normovolemic hemodilution.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2018-06 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Serum-Hematocrit | Postoperative 2 hour
  intergroup-difference immediately after surgery, %

SECONDARY OUTCOMES:
Serum-Ferritin level | Postoperative 2 hour
  intergroup-difference in postoperative hematocrit level, %
Changes of serum-Ferritin level | Postoperative 2 hour
  Intragroup-difference in the s-ferritin before and immediately after surgery, mg/dl
Transfusion amount | Postoperative 2 hour
  intergroup-difference in the amount of packed RBC transfused during surgery, unit

IPD SHARING:
Plan to Share IPD: No